CLINICAL TRIAL: NCT03438240
Title: Adding Dexmedetomidine Versus Fentanyl to Bupivacaine for Epidural Analgesia in Combination With General Anesthesia for Elective Lumbar Disc Operations: Prospective, Randomized Double-blinded Study
Brief Title: Dexmedetomidine Versus Fentanyl Plus Bupivacaine for Epidural Analgesia With General Anesthesia for Lumbar Disc Operations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R8 /2018
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-02

CONDITIONS: Anesthesia
MeSH Terms: interventions — Bupivacaine; Anesthetics, Local; Fentanyl; Analgesics, Opioid; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group BF (Active Comparator): Bupivacaine plus Fentanyl
  Interventions: Drug: Bupivacaine; Drug: Fentanyl
- Group BD (Active Comparator): Bupivacaine plus Dexmedetomidine
  Interventions: Drug: Bupivacaine; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine — patients will receive combined general anesthesia / epidural analgesia with 15 ml bupivacaine 0.20%
  Other Names: Local anesthetic
Drug: Fentanyl — Plus 50 µg fentanyl
  Other Names: Opioid
  Arms: Group BF
Drug: Dexmedetomidine — Plus 50 µg dexmedetomidine
  Other Names: alpha 2 sympathomimetic
  Arms: Group BD

SUMMARY:
The purpose of this study is to compare addition of dexmedetomidine or fentanyl to bupivacaine for epidural analgesia in combination with general anesthesia in elective lumbar spine operations as regard hemodynamic stability, postoperative pain control and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Physical status American Society of Anesthesiologist (ASA) I or II.
* First time elective lumbar dicsectomy or laminectomy

Exclusion Criteria:

* Patients who refuse to participate
* Body mass index (BMI) > 30
* Need an emergency lumbar disc operation
* ASA physical status > II
* Major illnesses (e.g. cardiac, respiratory, renal, liver)
* Coagulation abnormalities
* Hypovolemia
* History of increased intracranial pressure
* Convulsions
* Spinal stenosis
* Infection at needle insertion site
* Other contraindications to epidural procedure
* Allergy or contraindications to the drugs used in the study
* History of addiction or alcohol abuse
* Psychiatric illness or mental retardation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
First time to analgesic requirement | First 24 hours postoperatively
  After extubation, an intravenous patient-controlled analgesia system, will be connected to the patient (Accufuser Plus® 100 ml, Woo Young Medical Co, Korea) will be prepared with 60 ml normal saline containing 60 mg morphine, it will be programmed to give and 0.5 ml bolus dose with lockout interval of 8 minutes. Time to first Bolus will be estimated considering extubation time is the zero time.

SECONDARY OUTCOMES:
Total opioid consumption | First 24 hours postoperatively
  Total morphine consumption per twenty four hours will be estimated
Visual analogue scale (VAS) | First 24 hours postoperatively
  Pain scores will be evaluated by a blinded observer anesthesiologist at the time of arrival in the PACU, and 10, 20, 30 minutes, 1 h, 2h, 4, 6, 8, 10, 12, 16 and 24 hr thereafter using visual analogue scale (VAS) (0-10 cm: 0 = no pain, 10 = the worst pain possible). The patients will be instructed about usage of VAS preoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided